CLINICAL TRIAL: NCT06562556
Title: Impact of Breather Device on Ventilatory Effort in Patient With Myogenic Temporomandibular Joint Disorders
Brief Title: Impact of Breather Device on Ventilatory Effort in Patient With MTMD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Weaam Soliman Hassaneen, asssisstant lectruer, Misr University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: breather device for MTMD
Record Dates: First submitted 2024-08-13; First posted 2024-08-20 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: TMD

STUDY DESIGN:
Intervention Model Description: Group A: (Experimental group) Thirty patients, will receive a combined treatment program containing respiratory muscle training by the breather device with a conventional exercise program for MTMD for four consecutive weeks (3 sessions/ week). Group B: (Control group) Thirty patients, who will receive a conventional exercise program for MTMD for four consecutive weeks (3 sessions/ week)
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participant Group/Arm (Experimental): rThirty patients, will receive a combined treatment program containing respiratory muscle training by the breather device with a conventional exercise program for MTMD for four consecutive weeks (3 sessions/ week)
  Interventions: Device: the breather device; Other: conventional exercise program
- Control group/Arm (Other): Thirty patients, who will receive a conventional exercise program for MTMD for four consecutive weeks (3 sessions/ week).
  Interventions: Other: conventional exercise program

INTERVENTIONS:
Device: the breather device — investigate the effect of the breather device on ventilatory effort and in patients with myogenic temporomandibular joint disorders
  Arms: Participant Group/Arm
Other: conventional exercise program — -Therapeutic Ultrasound (US): Ultrasound therapy will be applied at the site of pain over the TMJ area with Frequency: 1 MHz, Mode: continuous, Duration: 6 min. each session 2-Myofascial release for masticatory muscles 3-The self-exercise Self exercise: include simplified myo-functional therapy. 10 repetitions, three: five times per day 4-Techniques to correct deglutition: swallowing a small amount of water and speaking while holding a semi-hard small object between the dental arches 5-Relaxation exercise of Masticator Muscle:10 repetitions, three.
  6-Strain-counterstain (SCS): applied on the tender or trigger points of neck muscles on improving pain and pressure pain sensitivity in neck muscles

SUMMARY:
PURPOSE:

The purpose of the study is to investigate the effect of the breather device on ventilatory effort and in patients with myogenic temporomandibular joint disorders To investigate the effect of the breather device on craniocervical angle and oral Health quality in patients with myogenic temporomandibular joint disorders

BACKGROUND:

TMDs affect between 5% and 12% of the population which is presented by symptoms such as pain in the masticatory muscles with a decrease in the mandible's movement. Other symptoms include ear pain, headache, joint sounds with mandible movement, and/or functional limitations in the jaw like swallowing difficulties commonly found. (Hatice ., et al 2023) Increased prevalence of TMDs has been linked to physical, psychological, and hormonal changes throughout pubertal development. The age predisposes to the development of masticatory system problems in students since symptoms peak between the ages of 20 and 40 years. Women of breeding age are the majority of TMD sufferers. The prevalence of TMD increases globally throughout adolescence and may vary from 7% to 30% of the population (Loster ., et al2017). Alterations of body posture, upper thoracic breathing pattern, and mouth breathing constitute causal factors for the overuse of the accessory inspiratory musculature, which generates hyperactivity and consequently, alteration of head position, and mandibular traction. (Kim., et al 2017)

HYPOTHESES:

There will be no significant effect of the breather device on ventilatory effort in patients with myogenic temporomandibular joint disorders.

There will be no significant effect of the breather device on a craniocervical angle and oral Health quality in patients with myogenic temporomandibular joint disorders RESEARCH QUESTION: Does the breather device can improve ventilatory effort in patients with myogenic temporomandibular joint disorders?.

DETAILED DESCRIPTION:
Randomized controlled trial which will be conducted on sixty female patients with chronic pain myogenous TMD for more than three months will be included in our study., their ages will range from 20 to 30 years. They will be selected from students of Misr University for Science and Technology to be enrolled in this study. They will participate in this study for 4 weeks The patients will participate and randomly be assigned into two equal groups. Group A: (Experimental group) Thirty patients, will receive a combined treatment program containing respiratory muscle training by the breather device with a conventional exercise program for MTMD for four consecutive weeks (3 sessions/ week).

Group B: (Control group) Thirty patients, who will receive a conventional exercise program for MTMD for four consecutive weeks (3 sessions/ week)

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:

  1. Sixty female patients who fulfilled the RDC/TMD criteria of myofascial pain and the presence of parafunctional habits, such as bruxism, teeth grinding, mouth breathing, and lip biting.
  2. The Patient's ages will range from 20 to 40 years.

  4- Patients with a waist-height ratio measuring less than 0.5. 5- Patients with a craniocervical angle measuring from 30 to 50° (Bo-Been et al., 2016).

  6- the patients have points from 20-65 on the Fonseca Anamnestic Index (FAI) 7- the patients have the willingness to participate in this study. 8- All patients will sign a consent form before starting the study.

Exclusion Criteria:

Patients will meet one of the following criteria will be excluded from the study:

1. patients undergo surgery or trauma in the orofacial region; systemic or degenerative odontologic disease.
2. The patient has Surgery or trauma in the spine and upper limb.
3. Patients suffering from rheumatic diseases and other severe comorbidities.
4. Patients suffering from any respiratory diseases (restrictive, obstructive, suppurative diseases).
5. Patients suffering from neurological disorders affecting respiratory muscles or any muscular dystrophies

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — sixty women patients with chronic pain myogenous TMD for more than three months will be included in our study., their ages will range from 20 to 40 years. They will be selected from students of Misr University for Science and Technology to be enrolled in this study. They will participate in this study for 4 weeks.
Enrollment: 60 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
spirometer | 4 weeks
  measure ventilatory function test in percentage
  1. Forced expiratory volume in the first second (FEV1)
  2. Forced vital capacity (FVC).
  3. FEV1/FVC ratio.
  4. Maximal Ventilator Volume (MVV)
Surface electromyography (sEMG): | 4 weeks
  To evaluate nerve-muscle activity during static conditions and active movements of the scalene muscle and sternocleidomastoid muscle

SECONDARY OUTCOMES:
Fonseca Anamnestic Index (FAI) | 4 weeks
  to diagnose TMD and evaluate the severity of the disorder. FAI is a functional assessment scale, which contains 10 objective questions which there are three possible answers: no 0 points, sometimes 5 points, and yes 10 points. The total score gives the FAI classification as follows: 70-100 points, severe TMD. 45-65 points, moderate TMD. 20-40 points, mild TMD. 0-15 points, TMD-free. TMD is diagnosed on FAI scores of ≥20
Numeric Pain Rating Scale (NPRS) | 4 weeks
  To assess neck Pain intensity on a scale from 0 to 10 using whole Arabic numbers.
craniocervical angle measuring | 4 weeks
  Kinovea software
The Oral Health Impact Profile Questionnaire OHIP-14 | 4 weeks
  to determine oral health quality. comprises 14 items that explore seven dimensions of impact: functional limitation, physical pain, psychological discomfort, physical disability, psychological disability, social disability, and handicap. The responses were classified using the Likert scale with five options ranging from "never" (0) to "very often" (4)
Tape Measurement tool and height scale | preassessment
  To measure the waist/ height ratio

REFERENCES:
- [Result] Walczynska-Dragon K, Baron S, Nitecka-Buchta A, Tkacz E. Correlation between TMD and cervical spine pain and mobility: is the whole body balance TMJ related? Biomed Res Int. 2014;2014:582414. doi: 10.1155/2014/582414. Epub 2014 Jun 19. PMID 25050363